CLINICAL TRIAL: NCT02615678
Title: Acupuncture for Chemotherapy-Induced Peripheral Neuropathy in Breast Cancer Patients- A Case Series
Brief Title: Acupuncture for CIPN in Breast Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Southern California University of Health Sciences (Other)
Responsible Party: Principal Investigator, Sivarama Vinjamury, Professor, Southern California University of Health Sciences
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VINJ007
Record Dates: First submitted 2015-11-21; First posted 2015-11-26 (Estimated); Last update posted 2019-05-16 (Actual); Status verified 2019-05

CONDITIONS: Sensation Disorders; Neuropathy
Keywords: neuropathy; peripheral; chemotherapy; breast cancer
MeSH Terms: conditions — Sensation Disorders; Breast Neoplasms | interventions — Acupuncture Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Acupuncture (Experimental): Acupuncture including scalp needling will be applied to selected points based on literature
  Interventions: Device: Acupuncture

INTERVENTIONS:
Device: Acupuncture — Acupuncture twice a week for 6 weeks then one treatment a week for 4 weeks. Total 16 treatments in 10 weeks.

SUMMARY:
The aim of this study is to collect preliminary data on the effectiveness of acupuncture for the treatment of CIPN in breast cancer patients.

DETAILED DESCRIPTION:
Ideally 10 patients experiencing peripheral neuropathy due to chemotherapy from breast cancer treatment will be included in this study.They will receive 16 total acupuncture treatments over 10 weeks including various points based off of research and classical text and scalp acupuncture.

ELIGIBILITY:
Inclusion criteria:

1. Minimum of 18 years of age
2. Currently receiving neurotoxic chemotherapy
3. Experiencing symptoms of chemotherapy induced neuropathy for at least 1 month
4. Have a minimum score of 3 on the VAS should have a grade II CIPN on NCICTC
5. Willing to sign an informed consent
6. Stable treatment for more than two months before screening

   * Stable treatment is defined as no change in the type and dose of medications 2 months prior to enrollment.
   * Once enrolled, the patients will be asked to remain on the same type and dose of the medications for neuropathy

Exclusion Criteria:

1. Receiving any treatment to prevent neuropathy 2 weeks prior to the screening
2. Pre-existing peripheral neuropathy due to any other cause than chemotherapy
3. Pre-existing conditions like pregnancy, uncontrolled diabetes, hypertension, cardiovascular disorders, bleeding disorders, depression (BDI > 21)
4. Unwilling to follow the protocol
5. Individuals who are receiving government disability assistance

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2015-10; Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Changes in perceived neuropathy as measured by EORTC CIPN-20 | At baseline, week 6 (treatment 12) and at week 10 (treatment 16)
  This is a 20-item self-report multidimensional CIPN specific scale that measures sensory, motor and autonomic symptoms of a 1-4 Likert scale.

SECONDARY OUTCOMES:
Changes in perceived neuropathy as measured by Functional Assessment of Cancer Therapy/Gynecologic Oncology Group-Neurotoxicity (FACT-GOG) Questionnaire | At baseline, week 6 (treatment 12) and at week 10 (treatment 16)
Changes in perceived neuropathy as measured by Visual Analogue Scale of Pain | At baseline, week 6 (treatment 12) and at week 10 (treatment 16)
Changes in quality of life as measured by EORTC QLQ-30 | At baseline, week 6 (treatment 12) and at week 10 (treatment 16)

CONTACTS AND LOCATIONS:
Overall Officials: Sivarama Vinjamury, MD, MAOM, Principal Investigator — Southern California University of Health Sciences, College of Eastern Medicine
Locations (1):
- Southern California University of Health Sciences, Whittier, California, United States